CLINICAL TRIAL: NCT02907840
Title: Prediction of Response to Recruitment Maneuvers in Patients With Acute Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Researcher, Università degli Studi di Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 141285
Record Dates: First submitted 2016-09-05; First posted 2016-09-20 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recruitment (Experimental): Lung aeration monitored by Swisstom BB2 during PEEP steps and recruitment maneuver
  Interventions: Device: Swisstom BB2

INTERVENTIONS:
Device: Swisstom BB2 — Electrical impedance tomography lung monitoring uses a dedicated belt placed around patient's thorax to detect change in impedance due to change in aeration within the thorax

SUMMARY:
The study will explore the possibility to predict potential for recruitment in acute hypoxemic respiratory failure patients by electrical impedance tomography (EIT) Swisstom BB2 (Swisstom, Landquart, Switzerland) during stepwise increase in positive end-expiratory pressure (PEEP) followed by recruitment maneuver (RM). It will compare data obtained by EIT to those obtained by pressure-volume (P-V) curves on respiratory system mechanics and data on pulmonary gas exchange.

DETAILED DESCRIPTION:
The investigators will monitor lung ventilation by EIT during the whole protocol and perform P-V curves and arterial blood gas analysis at every step of the protocol.

Participants will be sedated and paralyzed, ventilated in volume-controlled with protective ventilation (tidal volume=6-8 mL/Kg of predicted body weight and respiratory rate set to obtain normal pH) then the protocol will follow 5 steps each lasting 20 minutes to obtain clinical stability:

1. PEEP 5 centimeter of water (cmH2O)
2. PEEP 10 cmH2O
3. Recruitment maneuver followed by PEEP 15 cmH2O
4. PEEP 10 cmH2O
5. PEEP 5 cmH2O

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute hypoxemic respiratory failure defined by recent known clinical insult or worsening of respiratory symptoms and arterial pressure of oxygen to inspired fraction of oxygen ratio (PaO2/FiO2) ≤300 mmHg
* Patient on invasive mechanical ventilation
* Age ≥18 years
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Unstable hemodynamic condition requiring blood transfusion or adjustment of inotropics more often than every hour
* FiO2 ≥80% or clinical suspicion of pulmonary embolism
* Pneumothorax
* Chronic obstructive pulmonary disease (COPD) with clinical symptoms of lung emphysema as evidenced by chest radiography or computed tomography or autoPEEP > 5 cmH2O
* Intracranial hypertension
* Impossibility to correctly position the EIT belt (e.g., dressings, chest drainage, etc.)
* Contraindications to EIT (e.g., implantable cardiac defibrillator, pacemaker, instable spinal lesions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Significant reduction in silent spaces (i.e. non ventilated lung areas) during incremental PEEP steps | Within 20 minutes from PEEP increase

CONTACTS AND LOCATIONS:
Overall Officials: Savino Spadaro, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Azienda Ospedaliero Universitaria Sant'Anna, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scaramuzzo G, Spadaro S, Waldmann AD, Bohm SH, Ragazzi R, Marangoni E, Alvisi V, Spinelli E, Mauri T, Volta CA. Heterogeneity of regional inflection points from pressure-volume curves assessed by electrical impedance tomography. Crit Care. 2019 Apr 16;23(1):119. doi: 10.1186/s13054-019-2417-6. PMID 30992054
- [Derived] Spadaro S, Mauri T, Bohm SH, Scaramuzzo G, Turrini C, Waldmann AD, Ragazzi R, Pesenti A, Volta CA. Variation of poorly ventilated lung units (silent spaces) measured by electrical impedance tomography to dynamically assess recruitment. Crit Care. 2018 Jan 31;22(1):26. doi: 10.1186/s13054-017-1931-7. PMID 29386048